CLINICAL TRIAL: NCT04359719
Title: The Comparison Between Free Thyroxine and Thyroid Stimulating Hormone Levels on Melasma Severity: A Cross Sectional Study
Brief Title: Comparison Between Free Thyroxine and Thyroid Stimulating Hormone Levels on Melasma Severity
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD-Head of Division of Cosmetic Dermatology, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Other Study IDs: ThyrMel
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Melasma
Keywords: mMASI; Janus II facial analysis system; TSH; FT4
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group mild melasma: This subjects according to the modified melasma area and severity index (mMASI) score. Variables that are measure by mMASI scoring includes the degree of darkness and involvement of area. Darkness component is used to replace pigmentation and intensity in MASI scoring with modification (mMASI). Assessment using mMASI is highly dependent on the operator; hence, a new objective examination to assess skin pigmentation have been developed, which is the facial imaging analysis.
  The level of serum FT4 and TSH were then measured in both groups of the patients. In addition, the degree of skin pigmentation was also measured by using the Janus II facial analysis system. In this study, there were two modalities used in the Janus II facial analysis system, which is the polarization light and ultraviolet light.
  In addition, this study also analyzes the level of serum FT4 and TSH with the result of Janus II facial analysis system scoring.
- Group Moderate-severe melasma: This subjects according to the modified melasma area and severity index (mMASI) score. Variables that are measure by mMASI scoring includes the degree of darkness and involvement of area. Darkness component is used to replace pigmentation and intensity in MASI scoring with modification (mMASI). Assessment using mMASI is highly dependent on the operator; hence, a new objective examination to assess skin pigmentation have been developed, which is the facial imaging analysis.
  The level of serum FT4 and TSH were then measured in both groups of the patients. In addition, the degree of skin pigmentation was also measured by using the Janus II facial analysis system. In this study, there were two modalities used in the Janus II facial analysis system, which is the polarization light and ultraviolet light.
  In addition, this study also analyzes the level of serum FT4 and TSH with the result of Janus II facial analysis system scoring.

SUMMARY:
The objective of the study was to compare the level of serum FT4 and TSH in patients with mild melasma and moderate-severe melasma. The determination of melasma lesion could also be known by using Janus II facial analysis UV light and polarization light to analyze the pattern of hyperpigmentation on melasma. This was a descriptive-analytic study used a cross-sectional method that was performed in 2019 at two different dermatology and venerology clinics in Indonesia, Cipto Mangunkusumo Hospital Jakarta and Gatot Subroto Army Hospital Jakarta. Forty-eight subjects with melasma, 50% diagnosed with mild melasma and 50% with moderate-severe melasma according to the modified melasma area and severity index (mMASI) score. The level of serum FT4 and TSH were then measured in both groups of the patients.

DETAILED DESCRIPTION:
Melasma has been suspected to be linked with thyroid hormone. There is no study that explains the association of thyroid hormone level with melasma severity.

This study aims to find the difference in the levels of thyroid hormone in varying severity of melasma.

This was a descriptive-analytic study used a cross-sectional method that was performed in 2019 at two different dermatology and venerology clinics in Indonesia, Cipto Mangunkusumo Hospital Jakarta and Gatot Subroto Army Hospital Jakarta.

Forty eight patients participated in this study, 50% diagnosed with mild melasma and 50% with moderate-severe melasma. Subjects are chosen consecutively based on mMASI and Janus II measurement. The level of serum FT4 and TSH were then measured in both groups of the patients. The data is tabulated and a comparative analysis of serum FT4 and TSH levels with mild and moderate-severe melasma is done. In addition, this study also analyzes the level of serum FT4 and TSH with the result of Janus II facial analysis system scoring. The same method of analysis was done to know the association between mMASI and examination by using Janus II facial analysis system.

This study aims to find the difference in the levels of thyroid hormone in varying severity of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years
* Melasma lesions on the facial area.
* Willing to be the subject of research and sign a letter of research approval after being given an explanation (informed consent)

Exclusion Criteria:

* Pregnancy
* History of thyroid disease
* Using drugs that can affect the thyroid (glucocorticoids, lithium, amiodarone, iodide, octreotide)
* Using hormonal contraception for the past 1 year
* Using anti-seizure drugs
* Using hormone replacement therapy (HRT)
* Brown spots on the face preceded by reddish spots
* Brown spots on the face preceded by contact with facial whitening ingredients (hydroquinone)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population is patients with melasma in Indonesia aged 20-50 years.
  Affordable population are patients with melasma who come to the Skin and Genital Clinic of RSCM aged 20-50 years in the study period.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
association of serum TSH and FT4 level with the severity degree of melasma | 2 weeks: 15 - 26 July 2019
  There are no association between the level of serum TSH and FT4 and various degrees of melasma

SECONDARY OUTCOMES:
The correlation of serum TSH and FT4 levels with the Janus facial analysis system | 2 weeks: 15 - 26 July 2019
  The correlation is only found between the level of serum FT4 and Janus polarization test

OTHER OUTCOMES:
Correlation between Janus II facial analysis system and mMASI score in the mMASI darkness score assesment | 2 weeks: 15 - 26 July 2019
  A weak positive correlation is found between mMASI score and Janus II facial analysis system with polarization light test. Meanwhile, there is no correlation found between the Janus UV test and mMASI darkness score.

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Irma B Sitohang, MD, PhD, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No